CLINICAL TRIAL: NCT05126069
Title: Longitudinal Gelatin Stent vs. Trabeculectomy (LongGVT Study): Ab Interno Gelatin Stent With Mitomycin C Versus Trabeculectomy With Mitomycin C: a Retrospective Cohort Analysis
Brief Title: Ab Interno Gelatin Microstent With MMC vs. Trabeculectomy With MMC: 3 Year Retrospective Cohort Analysis
Acronym: LongGVT
Status: Completed | Type: Observational
Sponsor: Prism Eye Institute (Other)
Responsible Party: Principal Investigator, Iqbal Ahmed, Chief Innovation Officer, Prism Eye Institute
Other Study IDs: 2018-10376
Record Dates: First submitted 2021-11-05; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Filtering Surgery; Trabeculectomy
Keywords: Xen; Ab Interno Gelatin Microstent
MeSH Terms: interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Standalone Xen45: consecutive patients from June 2012 - July 2017 who received standalone Xen45®
  Interventions: Device: Ab interno gelatin microstent
- Standalone Trabeculectomy: consecutive patients from June 2012 - July 2017 who received standalone trabeculectomy
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: Ab interno gelatin microstent — Ab interno gelatin microstent
  Groups: Standalone Xen45
Procedure: Trabeculectomy — Trabeculectomy
  Groups: Standalone Trabeculectomy

SUMMARY:
To compare 3-year post-operative efficacy and safety of standalone ab interno gelatin microstent (Xen45®) versus trabeculectomy.

DETAILED DESCRIPTION:
This is a single-center retrospective cohort study. Patients included were consecutive patients from June 2012 - July 2017 who received standalone Xen45® or standalone trabeculectomy. The primary outcome was time to failure, defined as intraocular pressure (IOP) outside of 6mmHg - 17mmHg on no medications on two consecutive visits despite in-clinic maneuvers (including needling). Secondary outcomes included IOP cutoffs of 14mmHg and 21mmHg with and without medications, as well as interventions, complications, and reoperations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-90
* primary or pigmentary/pseudoexfoliative open angle, primary closed angle, narrow angle or combined mechanism glaucoma
* IOP of 18-40 on maximum tolerated medical therapy
* received a gelatin stent 45 with MMC or a trabeculectomy with MMC at Prism Eye Institute from June 2012 to July 2018, and have at least 3 years of follow-up.

Exclusion Criteria:

* Other forms of glaucoma
* prior incisional glaucoma surgery
* CPC
* combined surgery (cataract, cornea, or retina)
* prior corneal graft (PKP, DALK, DSAEK, DMEK)

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients who received received a gelatin stent 45 with MMC (mitomycin C) or a trabeculectomy with MMC
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
time to failure | up to 3 years
  defined as intraocular pressure (IOP) outside of 6mmHg - 17mmHg on no medications on two consecutive visits despite in-clinic maneuvers (including needling)

SECONDARY OUTCOMES:
included IOP cutoffs of 14mmHg and 21mmHg with and without medications, as well as interventions, complications, and reoperations | up to 3 years
  Secondary outcomes included IOP cutoffs of 14mmHg and 21mmHg with and without medications, as well as interventions, complications, and reoperations.

CONTACTS AND LOCATIONS:
Locations (1):
- Prism Eye Institute, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] J Liu, M Schlenker, I Ahmed. Long-Term Efficacy & Safety of Standalone Ab Interno Gelatin Microstent Implantation with MMC Vs. Trabeculectomy with MMC: 3 Year Follow-up. ASCRS Conference 2021.
- See also: Related Info — https://ascrs.org/clinical-education/abstracts/2021/longterm-efficacy--safety-of-standalone-ab-interno-gelatin-microstent-implantation-with-mmc-vs-trabe